CLINICAL TRIAL: NCT06821607
Title: Telerehabilitation for Patients With Chronic Low Back Pain (TeleBACK Clinical Trial)
Acronym: TeleBACK
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: University of Utah (Other); Intermountain Health Care, Inc. (Other); Patient-Centered Outcomes Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB00460142
Record Dates: First submitted 2025-02-06; First posted 2025-02-12 (Actual); Last update posted 2025-04-10 (Actual); Status verified 2025-04

CONDITIONS: Chronic Low Back Pain
Keywords: chronic low back pain; physical therapy; telehealth; telerehabilitation
MeSH Terms: interventions — Telerehabilitation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- In-Clinic Physical Therapy (Active Comparator): Patients in this group will receive all PT sessions in-clinic with a trained physical therapist. Treatment provided for this group will be consistent with evidence-based guidelines that recommend patient education, exercise instruction, manual therapy interventions, and psychosocial interventions. Specific interventions to be provided within each of these categories: Education, Exercise, Manual Therapy, and Psychosocial interventions. Components of the intervention will be determined by the treating therapist based on patients' symptoms, examination findings, and patients' preferences and goals.
  Interventions: Behavioral: In-Clinic Physical Therapy
- Telehealth Physical Therapy (Telerehabilitation) (Experimental): Those randomized to telerehabilitation will receive all PT care, including the initial evaluation and 7 follow-up sessions, via real-time video conferencing technology. Like the interventions provided to those receiving in-clinic PT, treatments provided in the telerehabilitation group will be consistent with evidence-based guidelines, adapted for delivery via real-time video visits. Consistent with the in-clinic group, specific interventions will be selected by the treating physical therapist based on patients' symptoms, examination findings, and preferences and goals.
  There will be an emphasis: Open-ended questions to allow patients to describe impairments and limitations; Review patient-reported measures of disability and pain intensity to help identify functional impairments; and Clinical examination of spinal movements and impairments in strength, flexibility, and joint mobility.
  Interventions: Behavioral: Telehealth Physical Therapy (Telerehabilitation)

INTERVENTIONS:
Behavioral: In-Clinic Physical Therapy — Patients in this group will receive all PT sessions in-clinic with a trained physical therapist. Treatment provided for this group will be consistent with evidence-based guidelines that recommend patient education, exercise instruction, manual therapy interventions, and psychosocial interventions. Specific interventions to be provided within each of these categories: Education, Exercise, Manual Therapy, and Psychosocial interventions. Components of the intervention will be determined by the treating therapist based on patients' symptoms, examination findings, and patients' preferences and goals.
  Arms: In-Clinic Physical Therapy
Behavioral: Telehealth Physical Therapy (Telerehabilitation) — Those randomized to telerehabilitation will receive all PT care, including the initial evaluation and 7 follow-up sessions, via real-time video conferencing technology. Like the interventions provided to those receiving in-clinic PT, treatments provided in the telerehabilitation group will be consistent with evidence-based guidelines, adapted for delivery via real-time video visits. Consistent with the in-clinic group, specific interventions will be selected by the treating physical therapist based on patients' symptoms, examination findings, and preferences and goals. There will be an emphasis: Open-ended questions to allow patients to describe the participant's impairments and limitations; Review patient-reported measures of disability and pain intensity to help identify functional impairments; and Clinical examination of spinal movements and impairments in strength, flexibility, and joint mobility.
  Arms: Telehealth Physical Therapy (Telerehabilitation)

SUMMARY:
The investigators will conduct a prospective, randomized, clinical trial addressing key questions to understanding the effectiveness of telerehabilitation (physical therapy delivered via video-visits) and in-clinic physical therapy for patients with chronic low back pain (LBP). The investigators also seek to understand how patients engage with both care options and how these treatment options influence other LBP-related healthcare utilization.

The investigators will explore implementation outcomes using a mixed methods approach consisting of electronic surveys and semi-structured interviews with patients, physical therapists, practice managers, and outpatient services administration focusing on perceived quality and impact on barriers to care. The investigators will enroll 1000 patients with chronic LBP seeking outpatient care at the healthcare systems in Maryland (Johns Hopkins Medicine (JHM)) and Utah (University of Utah (UU) and Intermountain Healthcare (IHC)). Eligible patients will provide informed consent and be randomized to receive telerehabilitation or in-clinic physical therapy delivered by a trained physical therapist. Primary effectiveness outcome is the difference in change in LBP-related disability (Oswestry Disability Index) after 8 weeks of treatment.

DETAILED DESCRIPTION:
Low back pain (LBP) is a nearly universal human experience with 80% of adults having at least one episode in the adult's lifetime and 25% of adults reporting LBP lasting at least 1 day in the past 3 months. Not only is LBP exceedingly common, but it can be very burdensome. The tremendous burden imposed by LBP on health and well-being was recently highlighted in the Global Burden of Disease initiative of the World Health Organization, showing that LBP is associated with greater disability and overall burden for affected individuals than depression, Alzheimer's disease, substance abuse disorders, or arthritis. This high ranking of LBP reflects the sheer number of people who experience the condition and the amount of pain, functional loss, and overall diminishment in quality of life that these individuals experience. It is not surprising that LBP imposes a substantial societal burden being the most common condition encountered in healthcare and the 3rd costliest medical condition, behind only diabetes and heart disease. Despite intensive and expensive treatment efforts, the number of individuals impacted by chronic LBP continues to increase. Ineffective LBP management by health care systems is also contributing to the crisis of opioid over-prescribing.

Physical therapy (PT) has been found to be effective in reducing pain and disability related to LBP and as such, is recommended as the first line of treatment for LBP in clinical practice guidelines. Studies have shown that providing timely access to PT leads to significant decreases in pain and disability compared to usual care and has been associated with decreased odds of receiving advanced imaging, injection, surgery, or opioids over the next year. Despite the benefits of PT, only 7-13% of patients with LBP receive PT services. This low rate of utilization is likely related to barriers surrounding access (i.e., wait times, cost) and logistics (i.e., missed work time, transportation), which have been reported as reasons for not attending PT in previous studies. While these barriers are not unique to PT, the frequency of PT visits (1-3 times per week) and the length of PT care (6-12 weeks) exacerbate already existing barriers to attending in-person visits. Importantly, these barriers are amplified among minority groups and those living in rural areas of the country - minority individuals are 26% less likely than non-minority individuals to receive PT services for musculoskeletal pain.

The COVID-19 pandemic has facilitated the rapid emergence of remotely-delivered PT (i.e., telerehabilitation). Prior to the pandemic, outpatient PT was delivered almost exclusively in-person. However, as the pandemic began, policy changes led to major expansions in the way that PT is delivered. In early 2020, the Center for Medicare and Medicaid Services (CMS) announced temporary authorization for reimbursement of PT services delivered using real-time video visits. Shortly afterwards, the majority of commercial payors followed suit. A non-randomized clinical trial was recently conducted that found that patients with chronic spine pain experienced similar changes in pain, disability and quality of life with multidisciplinary rehabilitation delivered using real-time video visits compared to those that received in-clinic care. A prospective longitudinal study conducted by the study team found that a standardized PT protocol delivered using real-time video visits resulted in significant improvement in disability, pain intensity, pain interference, physical function and sleep disturbance among patients with chronic LBP.

The investigators will compare the effectiveness of telerehabilitation and in-clinic PT for patients with chronic LBP to demonstrated that telerehabilitation will provide non-inferior clinical effects to in-clinic PT.

The investigators propose to enroll 1,000 patients with chronic LBP who present to primary or specialty care at one of three health systems in Baltimore and Utah. Patients will be randomly assigned to receive an 8-session evidence-based PT treatment delivered via in-person or telehealth visits and will be followed for 12 months. Primary outcomes will be disability. Secondary outcomes will be pain intensity and interference, physical function, and patient engagement with treatment. Exploratory outcomes will be mental health, fatigue, social participation, and opioid and other LBP-related healthcare utilization. Moderating factors will be psychosocial risk for poor outcome and pain self-efficacy. Results will provide important information for patients, clinicians, physical therapists, and payers to make informed decisions about optimizing delivery of evidence-based physical therapy to improve quality of life in patients with chronic LBP.

ELIGIBILITY:
Inclusion Criteria:

* Primary care visit in the past 90 days with an LBP-related ICD-10 diagnosis.
* At least moderate levels of pain and disability requiring Oswestry score ≥24% and average pain rating ≥ 4/10 points.
* Meets NIH Task Force2 definition of chronic LBP based on two questions: 1) How long has LBP has been an ongoing problem? and 2) How often has LBP been an ongoing problem over the past 6 months? A response of greater than 3 months to question 1, and "at least half the days in the past 6 months" to question 2 is required to satisfy the NIH definition of chronic LBP.
* Can speak and understand English or Spanish (Utah sites only).

Exclusion Criteria:

* Recent history (last 6 months) of lumbar spine surgery.
* Possible non-musculoskeletal cause for low back pain symptoms (e.g., pregnancy).
* Evidence of serious pathology as a cause of LBP including neoplasm, inflammatory disease (e.g., ankylosing spondylitis), vertebral osteomyelitis, etc.
* Neurological disorder resulting in severe movement disorder, or schizophrenia or other psychotic disorder.
* Knowingly pregnant

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 1000 (Estimated)
Dates: Start 2025-04-01 (Actual); Primary Completion 2029-09-30 (Estimated); Study Completion 2030-05-01 (Estimated)

PRIMARY OUTCOMES:
Change in Oswestry Disability Index | Change from baseline to 3 months after treatment initiation
  LBP-related disability. The total score range is [0, 100] with higher values representing greater pain-related disability.

SECONDARY OUTCOMES:
Opioid Use | Change from baseline to 3 months after treatment initiation
  Self-reported and/or Electronic Health Record (EHR) documented opioid use
Change in Patient-Reported Outcomes Measurement Information System (PROMIS-29) Physical Function | Change from baseline to 3-, 6-, and 12- months after treatment initiation
  Physical function. The total score range is [0, 100] with higher scores indicating better physical function.
Change in Patient-Reported Outcomes Measurement Information System (PROMIS-29) Physical Function by Gender | Change from baseline to 3-, 6-, and 12- months after treatment initiation
  Physical function. The total score range is [0, 100] with higher scores indicating better physical function.
Change in Patient-Reported Outcomes Measurement Information System (PROMIS-29) Physical Function by Age Group | Change from baseline to 3-, 6-, and 12- months after treatment initiation
  Physical function. The total score range is [0, 100] with higher scores indicating better physical function.
Change in Patient-Reported Outcomes Measurement Information System (PROMIS-29) Physical Function by Psychosocial Risk | Change from baseline to 3-, 6-, and 12- months after treatment initiation
  Physical function. The total score range is [0, 100] with higher scores indicating better physical function.
Change in PROMIS Preference Score (PROPr) | Change from baseline to 3-, 6-, and 12-months after treatment initiation
  Total score range is [0, 100] with higher scores indicating better outcome.
Change in PROMIS Preference Score (PROPr) by Gender | Change from baseline to 3-, 6-, and 12-months after treatment initiation
  Total score range is [0, 100] with higher scores indicating better outcome.
Change in PROMIS Preference Score (PROPr) by Age Group | Change from baseline to 3-, 6-, and 12-months after treatment initiation
  Total score range is [0, 100] with higher scores indicating better outcome.
Change in PROMIS Preference Score (PROPr) by Psychosocial Risk | Change from baseline to 3-, 6-, and 12-months after treatment initiation
  Total score range is [0, 100] with higher scores indicating better outcome.
Percent of participants using non-opioid LBP-Related Healthcare Use | Change from baseline to 3-, 6-, and 12- months after treatment initiation
  Non-opioid LBP-related healthcare use (e.g., physician office visit, imaging, surgery)
Percent of participants using non-opioid LBP-Related Healthcare Use by Gender | Change from baseline to 3-, 6-, and 12- months after treatment initiation
  Non-opioid LBP-related healthcare use (e.g., physician office visit, imaging, surgery)
Percent of participants using non-opioid LBP-Related Healthcare Use by Age Group | Change from baseline to 3-, 6-, and 12- months after treatment initiation
  Non-opioid LBP-related healthcare use (e.g., physician office visit, imaging, surgery)
Percent of participants using non-opioid LBP-Related Healthcare Use by Psychosocial Risk | Change from baseline to 3-, 6-, and 12- months after treatment initiation
  Non-opioid LBP-related healthcare use (e.g., physician office visit, imaging, surgery)

OTHER OUTCOMES:
Percent of patients approached who accept participation | At screening
  Implementation - Acceptability as assessed by percent of patients approached who accept participant
Percent of patients offered telerehabilitation | At screening
  Implementation - Adoption as assessed by percent of patients offered tele-rehabilitation
Percent of intervention sessions completed | 3 months after treatment initiation
  Implementation - Feasibility as assessed by percent of intervention sessions completed
Percent of core treatment components provided during intervention sessions | 3 months after treatment initiation
  Implementation - Fidelity as assessed by percent of core treatment components provided during intervention sessions

CONTACTS AND LOCATIONS:
Overall Officials: Richard L. Skolasky, Sc.D., Principal Investigator — Johns Hopkins University; Kevin McLaughlin, D.P.T., Principal Investigator — Johns Hopkins School of Medicine
Locations (3):
- United States (3):
  - Johns Hopkins University School of Medicine, Baltimore, Maryland
  - Intermountain Healthcare, Salt Lake City, Utah
  - University of Utah, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: Yes
The Research Team at the Johns Hopkins University for the proposal titled "Telerehabilitation for Patients with Chronic Low Back Pain (TeleBACK Clinical Trial) agree to accept the overall governance, common protocols, publication policies, collaborative procedures, confidentiality, and data sharing plans to be developed by the Patient-Centered Outcomes Research Institute (PCORI). The following document exists to reflect best practices for data acquisition, management, stewardship, and dissemination that are consistent with the PCORI Public Access and Data Sharing Policy.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data will be available after final dataset is closed, curated, and uploaded to the data sharing platform. Data will be available in perpetuity.
Access Criteria: Data will be accessible on a closed-access basis. Researchers will have to request access and have this request be approved.